CLINICAL TRIAL: NCT03182491
Title: Mechanisms of Anaphylaxis
Acronym: ANAMEK
Status: Active, not recruiting | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/1635
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Anaphylaxis; Allergy; Transfusion Reaction; Febrile Transfusion Reaction
Keywords: Platelet activating factor; Basophil activation test; Anaphylatoxins
MeSH Terms: conditions — Anaphylaxis; Hypersensitivity; Transfusion Reaction | interventions — Basophil Degranulation Test

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Biospecimen Retention: Samples With DNA — Serum samples, plasma samples, full blood-samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Anaphylaxis
  Interventions: Diagnostic Test: Biomarkers (platelet activating factor [PAF], anaphylatoxins) and basophil activation test (BAT)
- Febrile transfusion reactions
  Interventions: Diagnostic Test: Biomarkers (platelet activating factor [PAF], anaphylatoxins) and basophil activation test (BAT)
- Mild allergic reactions
  Interventions: Diagnostic Test: Biomarkers (platelet activating factor [PAF], anaphylatoxins) and basophil activation test (BAT)
- Healthy controls
  Interventions: Diagnostic Test: Biomarkers (platelet activating factor [PAF], anaphylatoxins) and basophil activation test (BAT)

INTERVENTIONS:
Diagnostic Test: Biomarkers (platelet activating factor [PAF], anaphylatoxins) and basophil activation test (BAT) — Analysis of biomarkers and basophil activation test

SUMMARY:
The purpose of this study is to explore different mechanisms for anaphylaxis and find novel biomarkers for this hypersensitivity syndrome. The study participants are patients with anaphylaxis, patients with mild allergic reactions, and patients with febrile transfusion reactions. The investigators will also include a group of healthy controls.

ELIGIBILITY:
Inclusion Criteria:

According to the specific cohort:

1. Diagnosis of anaphylaxis
2. Mild allergic reaction
3. Febrile transfusion reaction
4. Healthy, no known allergic disease

Exclusion Criteria:

Suspicion or diagnosed sepsis Children

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-04-28 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Clarify mechanisms for anaphylaxis and establish biomarkers for this syndrome | 2 days
  Immunological/nonimmunological mechanism

CONTACTS AND LOCATIONS:
Overall Officials: Torunn O Apelseth, MD, PhD, Study Director — Haukeland University Hospital; Morten Y Isaksen, MD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway